CLINICAL TRIAL: NCT00113919
Title: UARK 2003-25: A Phase I/II Open Label Study of IV Busulfan (Busulfex®) in Multiple Myeloma Patients Older Than 65 Years of Age or With Renal Insufficiency
Brief Title: UARK 2003-25: A Study of Intravenous (IV) Busulfan (Busulfex®) in Multiple Myeloma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-25
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Results first posted 2011-06-20 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma, MM
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Experimental): study-specific treatment: Busulfex according to study design: Level I 3.2 mg/kg over 6 hours x 2 days Level II 3.2 mg/kg over 6 hours x 3 days Level III 3.2 mg/kg over 6 hours x 4 days Level IV 4.3 mg/kg over 6 hours x 3 days Level V 5.6 mg/kg over 6 hours x 2 days Level VI 6.4 mg/kg over 6 hours x 2 days
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — Dexamethasone 40 mg PO 1-4 Thalidomide 200 mg PO 1-6 Cisplatin* 10 mg/m, Continuous infusion 1-4 Adriamycin** 10 mg/m2, Continuous infusion 1-4 Cyclophosphamide 400 mg/2, Continuous infusion 1-4 Etoposide 40 mg/m2, Continuous infusion 1-4 All doses will be based on calculated body weight (actual weight + ideal body weight ÷ 2) and height, and not to exceed a BSA of 2.0 m2 The daily dose of cyclophosphamide, etoposide, and cisplatin will be mixed in a 1L bag of NS to be UAMS infused over 24 hours. Adriamycin will be mixed in at least 50cc D5W to be infused over 24 hours
  Other Names: Busulfex

SUMMARY:
The purpose of this study is to find out if patients with high risk disease because of age or kidney status can be treated more safely with a drug called Busulfex® followed by autologous transplant compared to treatment with the standard drug called melphalan, which has been shown to be quite difficult to tolerate in patients with poor kidney function and patients over the age of 65 when given in high doses.

DETAILED DESCRIPTION:
This trial will determine the maximal dose of Busulfex® that can be given in a two, three, or four day period with acceptable toxicity to myeloma patients, who either are > or = 65 years of age or have renal insufficiency, defined as creatinine > 3g/dL or creatinine clearance < 30 ml/min.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have symptomatic multiple myeloma requiring treatment
* Patients must have been approved for single or tandem autologous transplant
* Patients must be > or = 65 years of age or diagnosed with renal insufficiency, defined as having a creatinine > 3 mg/dl or a creatinine clearance < 30 ml/minute
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted,
* Patients must have an ECHO or MUGA performed within 60 days prior to registration, LVEF > 40%.
* Bilirubin, SGOT, SGPT must be less than 1.5 times the upper limit of normal
* Patients must have evaluable myeloma marker for response such as: *Serum M protein >1g/dl or urine M protein >1g/24 hours and/or; *Bone marrow plasmacytosis with >20% plasma cells and/or; *Extramedullary plasmacytosis; *MRI/PET scan has focal lesions due to myeloma.
* Patients must be able to receive full doses of DT-PACE, in the opinion of the treating investigator, with the exception of cisplatin.
* Patients must have a performance status of 0-2 based on SWOG criteria unless the patient's status is due to active myeloma
* All patients must be informed of the investigational nature of the study and have signed an IRB-approved informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Serum transaminases > 1.5 x ULN and direct bilirubin > 1.5 mg/dl
* HIV positive or active Hepatitis B or Hepatitis C infection; (if serology is positive a quantitative PCR will be done).
* Patients with a prior malignancy in whom life expectancy is more likely to be determined by the prior malignancy than the myeloma. Patients must not currently be receiving therapy for the prior malignancy.
* Pregnant or nursing women. Women of childbearing potential must have a negative pregnancy test documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — UAMS
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Myeloma Institute for Research and Therapy, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a medical facility. The subjects were recruited from the physician's patient base.
Groups:
- Bisulfan: Bisulfan in Multiple Myeloma patients >65 years w/renal insufficiency
Period: Overall Study
Arm/Group | Bisulfan
Started | 14
Completed | 0
Not Completed | 14
Not completed — Physician Decision | 8
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Bisulfan
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximal Dose of Busulfex® Given in a 2, 3, or 4 Day Period With Acceptable Toxicity to Myeloma Patients
Description: maximal dose of Busulfex® that can be given in a two, three, or four day period with acceptable toxicity to myeloma patients, who either are > or = 65 years of age or have renal insufficiency, defined as creatinine > 3g/dL or creatinine clearance < 30 ml/min
Time Frame: three years
Arm/Group | Busulfex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Dependent on notification by patient. Once UAMS received notification, documentation submitted to IRB within one week.
Arm/Group | Bisulfan
Serious Adverse Events (participants affected / at risk) | 12/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bisulfan (N=14)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
acute respiratory distress due to fluid overload (General disorders) | 2 (2)
bacteremia (Infections and infestations) | 1 (1)
blood clot in Arteriovenous fistula (Blood and lymphatic system disorders) | 1 (1)
catheter related septecemia (General disorders) | 1 (1)
cholecystitis (General disorders) | 1 (1)
colitis, diarrhea (Gastrointestinal disorders) | 1 (1)
febrile neutropenia with hypotention (Cardiac disorders) | 1 (1)
fluid overload (General disorders) | 2 (2)
hypotension, edema and depression (General disorders) | 1 (1)
hypovolemic shock (General disorders) | 1 (1)
inflammation syndrome, cellulitis, pansinusitis (General disorders) | 1 (1)
nephrogenic fibrosing dermopathy (General disorders) | 1 (1)
pancytopenia (General disorders) | 1 (1)
renal failure (Gastrointestinal disorders) | 3 (3)
seizures (General disorders) | 2 (2)
septic shock (General disorders) | 1 (1)
shortness of breath and tachcardia (Cardiac disorders) | 1 (1)
staphylococcal infection (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination, only 5 of the 14 completed, reasons as follows:

Death Unrelated to Protocol Adverse Event Relapse Patient Choice

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes